CLINICAL TRIAL: NCT05563428
Title: Efficacy of Free Gingival Graft Versus Connective Tissue Graft in the Treatment of Gingival Recessions at the Lower Incisors: a RCT
Brief Title: Free Gingival Graft Versus Connective Tissue Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Isabelle Laleman, Chef de clinique, Centre Hospitalier Universitaire de Liege
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-242
Record Dates: First submitted 2022-09-21; First posted 2022-10-03 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Gingival Recession; Gingival Recession, Localized
Keywords: Gingival recession; Free gingival graft; Connective tissue graft
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Randomized, controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free gingival graft (Active Comparator): Free gingival graft will be conducted.
  Interventions: Procedure: Free gingival graft
- Connective tissue graft (Active Comparator): The recession will be treated with the pouch technique using a connective tissue graft.
  Interventions: Procedure: Connective tissue graft

INTERVENTIONS:
Procedure: Free gingival graft — A free gingival graft will be carried out for recession treatment.
  Arms: Free gingival graft
Procedure: Connective tissue graft — The pouch technique with a connective tissue graft will be carried out for recession treatment.
  Arms: Connective tissue graft

SUMMARY:
This study wil compare FGG and CTG for recession coverage in the anterior mandibula.

ELIGIBILITY:
Inclusion Criteria:

* ASA type I and II subjects
* Localized Gingival Recessions
* Recessions Cairo RT I-II-III
* FMPS < 10%
* FMBS< 10%
* <10 cigs/ day
* No contra-indication against oral surgical interventions
* Patient is able to give inform consent

Exclusion Criteria:

* Infection (local or systemic). Each infection will be evaluated prior to study procedure for suitability. Patients with gingivitis or local infection (fracture, apical reaction) will undergo a dental treatment prior to entering the study. In case of systemic infection, the evaluation will be based on medical anamneses, and if necessary will be referred to relevant medical tests.
* ASA type > II
* Current pregnancy or breastfeeding women
* Alcoholism or chronically drug abuse
* Smokers, ≳ 10 cigarettes per day
* Immunocompromised patients
* Uncontrolled diabetes
* Untreated periodontitis
* History of previous periodontal surgery (mucogingival or other) on the teeth to be included
* Presence of severe tooth malposition, rotation or significant version of the tooth to be treated
* Conditions or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of no-compliance or unreliability

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Digital mean root coverage | Baseline, 3 months, 6 months and up to 10 years after surgery
  Defined as the percentage of root coverage in the mid-buccal aspect, taking baseline as a reference. Measured by dividing the mean surface (in mm²) of the root covered by the procedure by the mean surface (in mm²) of root exposed at baseline.

OTHER OUTCOMES:
Complete root coverage | Baseline, 3 months, 6 months and up to 10 years after surgery
  Defined as the presence/absence of complete coverage of the recession at the mid-buccal aspect. It will be evaluated by taking the CEJ as a reference line, at the different timepoints.
Mean root coverage | Baseline, 3 months, 6 months and up to 10 years after surgery
  defined as the percentage of root coverage in the mid-buccal aspect, taking baseline as a reference. The MRC equals to the linear distance (in mm, using a probe) between the mid buccal point of the CEJ and the mid-buccal sulcus at baseline, divided by the distance between the mid buccal point of the CEJ and the mid buccal sulcus. The MRC will be measured as percentage (%)
Keratinized tissue height | Baseline, 3 months, 6 months and up to 10 years after surgery
  Defined as the linear height of keratinized tissue, measured between the mid-buccal sulcus of the treated tooth and the muco-gingival junction (in mm using a probe). It will be measured at baseline and at the different timepoints.
Recession reduction | Baseline, 3 months, 6 months and up to 10 years after surgery
  defined as the linear reduction in recession (in mm using a probe), at the mid buccal aspect, between baseline and the different timepoints.
Gingival thickness | Baseline, 3 months, 6 months and up to 10 years after surgery
  evaluated at baseline using couloured paperpoints inserted into the sulcus.
CAL | Baseline, 3 months, 6 months and up to 10 years after surgery
  defined as the change in Clinical Attachement of the gingival margin, measured linearly at the mid-buccal aspect, from the JEC to the bottom of the pocket, at the different timepoints.
PPD changes | Baseline, 3 months, 6 months and up to 10 years after surgery
  defined as the change in depth of the pocket, measured at the mid-buccal aspect using a probe, between baseline and the different timepoints. It will be measured at the different timepoints.
Dental hypersensitivity | Baseline, 3 months, 6 months and up to 10 years after surgery
  Assessed by 10 s air spray applied to the buccal cervical area (yes/no).
Root coverage esthetic score | Baseline, 3 months, 6 months and up to 10 years after surgery
  Evaluated at the different timepoints according to Cairo et al. (2009).
Biological complications reported by the investigators | Baseline, 3 months, 6 months and up to 10 years after surgery
  Biological complications reported by the investigators
Digital complete root coverage | Baseline, 3 months, 6 months and up to 10 years after surgery
  defined as the presence/absence of complete coverage of the recession at the mid-buccal aspect. It will be evaluated by taking the CEJ as a reference line, at the different timepoints, analyzed digitally
Digital recession reduction | Baseline, 3 months, 6 months and up to 10 years after surgery
  defined as the reduction in recession (in mm², measured digitally), at the mid buccal aspect, between baseline and the different timepoints. It will be measured at the different timepoints.
Digital Keratinized Tissue Height | Baseline, 3 months, 6 months and up to 10 years after surgery
  Defined as the changes in keratinized tissue surface (surface delimited mesio-distally by the perpendicular projection of a line passing by the contact-point and apico-coronally by the muco-gingival junction and the gingival margin, at the mid-buccal aspect of the tooth.
Digital gingival soft tissue profile | Baseline, 3 months, 6 months and up to 10 years after surgery
  Defined as the change in gingival soft tissue thickness between baseline and the different timepoints, measured at the mid buccal aspect, between baseline and the different timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Szoted Gilles, MSc, Principal Investigator — ULiège
Locations (1):
- CHU de Liège, Liège, Belgium